CLINICAL TRIAL: NCT00783276
Title: An fMRI Study of SYN115 in Cocaine Dependent Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DA009262-14; P50DA009262 (NIH); DPMCDA
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2016-07

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — tozadenant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Drug: PLACEBO
- SYN115 (Active Comparator)
  Interventions: Drug: SYN115

INTERVENTIONS:
Drug: SYN115 — 100 mg single dose
  Arms: SYN115
Drug: PLACEBO — PLACEBO
  Arms: Sugar Pill

SUMMARY:
The dopamine system is critical in modulation of reward and has been implicated in the initiation and maintenance of addiction (Volkow et al 2004). Medications that increase dopamine either directly or indirectly have been shown to have preliminary efficacy at reducing cocaine use in cocaine dependent subjects (Grabowski et al 2004a; Schmitz et al 2008). A novel class of medications that has recently been shown to indirectly modulate dopamine function is adenosine A2A receptor antagonists (Fuxe et al 2007). Based on their effect on dopamine function it has been suggested that these compounds may be efficacious in the treatment of drug addiction (Ferre et al 2007c). Before clinical efficacy studies are undertaken, more basic research on the effects of adenosine A2A antagonists on brain function and behavior are warranted. The aim of this study is to examine the acute effects of a single dose of the selective adenosine A2A antagonist (SYN115, Synosia Therapeutics, Chemical name: 4-Hydroxy-4-methyl-piperidine-1-carboxylic acid-(4-methoxy-7-morpholin-4-yl-benzothiazol-2-yl)-amide) on brain function and behavior in cocaine dependent individuals using functional magnetic resonance imaging (fMRI). To examine the effect of a single dose of SYN115 on brain function and behavior in cocaine dependent subjects.

Hypotheses:

1. SYN115 100 mg will increase brain activation in the dorsolateral prefrontal cortex compared to placebo in cocaine dependent subjects performing a working memory task.
2. SYN115 100 mg will increase brain activation in the ventral striatum compared to placebo in cocaine dependent subjects performing a reversal learning task.
3. SYN115 100 mg will reduce brain activation in the anterior cingulate gyrus and amygdala compared to placebo in cocaine dependent subjects performing a cocaine-word Stroop task.

ELIGIBILITY:
INCLUSION CRITERIA: (1) 13 Male and 13 female subjects age 18 to 50 who currently meet DSM-IV criteria for cocaine dependence. (2) At least one cocaine positive urine during screening. (3) Female subjects: a negative pregnancy test.

EXCLUSION CRITERIA: (1) current or past DSM-IV Axis I disorder other than substance abuse/dependence (2) any significant non-psychiatric medical illness requiring ongoing medical treatment (3) any clinically significant abnormality on EKG (4) hypertension (5) cardiovascular disease (6) substance dependence other than cocaine, marijuana, or nicotine within the last 3 months. (7) Positive breath alcohol (8) Positive urine drug screen for drugs other than cocaine or THC at the time of behavioral testing (9) For female subjects: known pregnancy or a positive pregnancy test or current breast feeding (10) Diagnosis of Adult Attention Deficit Disorder as determined by: a) meeting DSM-IV criteria for childhood ADHD, b) currently has impairing ADHD symptoms, c) ADHD symptoms can not have remitted at any period since childhood (11) HIV positive (12) I.Q. below 70 (13) Use of medications which affect the central nervous system (CNS) or could interact with SYN115. (13) History of pacemaker or metal implants or welding or metal work without protective eyewear.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
fMRI Brain Activation | Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, M.D., Principal Investigator — UTHSC-Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Moeller FG, Steinberg JL, Lane SD, Kjome KL, Ma L, Ferre S, Schmitz JM, Green CE, Bandak SI, Renshaw PF, Kramer LA, Narayana PA. Increased Orbitofrontal Brain Activation after Administration of a Selective Adenosine A(2A) Antagonist in Cocaine Dependent Subjects. Front Psychiatry. 2012 May 28;3:44. doi: 10.3389/fpsyt.2012.00044. eCollection 2012. PMID 22654774
- [Result] Lane S, Green C, Steinberg J, Ma L, Schmitz J, Rathnayaka N, Bandak S, Ferre S, Moeller F. Cardiovascular and Subjective Effects of the Novel Adenosine A(2A) Receptor Antagonist SYN115 in Cocaine Dependent Individuals. J Addict Res Ther. 2012 Mar 28;S1:009. doi: 10.4172/2155-6105.S1-009. PMID 22905331